CLINICAL TRIAL: NCT00913666
Title: A Pilot Multi-Center, Open-Label, Assessor Blinded, Prospective Profiling Study in MS Subjects Treated With AVONEX®, MS Subjects Naïve to Treatment, and Healthy Control Subjects
Brief Title: Pharmacodynamic Study to Better Understand the Therapeutic Response and Immunomodulatory Effects of Avonex in Multiple Sclerosis (MS) Patients and Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: C-863
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (No Intervention): Healthy Volunteers
- Group 2 (Experimental): MS patients previously naïve to interferon therapy
  Interventions: Drug: Interferon beta-1a (Avonex)
- Group 3 (Experimental): MS patients on Interferon beta-1a treatment with no history of breakthrough disease (clinically stable)
  Interventions: Drug: Interferon beta-1a (Avonex)
- Group 4 (Experimental): MS patients on interferon beta-1a treatment with a history of breakthrough disease.
  Interventions: Drug: Interferon beta-1a (Avonex)

INTERVENTIONS:
Drug: Interferon beta-1a (Avonex) — 30 mcg by intramuscular injection once a week
  Other Names: Avonex
  Arms: Group 2; Group 3; Group 4

SUMMARY:
This study will look at differences in bioanalytical measures among different groups of MS patients and Healthy Volunteers, when administered interferon beta-1a.

ELIGIBILITY:
Inclusion Criteria:

Healthy Control Subjects (Group 1)

* Must be in general good health.
* Must not have received interferons in the past.

All MS Subjects

* Clinical or laboratory-supported diagnosis of relapsing remitting MS (McDonald et al, criteria numbers 1-4).
* Either on AVONEX® or treatment-naïve.
* Have an EDSS score between 0.0 and 5.5, inclusive.

Exclusion Criteria:

* History of severe allergic or anaphylactic reaction or hypersensitivity to human albumin, to any interferon, to other components of the drug formulation.
* History of intolerance to acetaminophen, ibuprofen, naproxen, and aspirin that would preclude the use of at least one of these during the study.
* History of any clinically significant (as determined by the investigator) cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease.
* History of malignancy.
* The presence of any significant medical condition or psychiatric illness not due to MS that, in the investigator's opinion, would interfere with therapy
* History of uncontrolled seizures within the 3 months prior to enrollment.
* History of suicidal ideation or an episode of severe depression within the 3 months prior to enrollment.
* Serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., pneumonia, septicemia) within 8 weeks prior to enrollment.
* Positive for human immunodeficiency virus (HIV), hepatitis C antibody (HCV) or positive for hepatitis B surface antigen (HbsAg) at screening.

Other inclusion and exclusion criteria apply as per protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2002-11; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Changes in bioanalytical measures after receiving therapy for 3 to 6 months | Study duration is 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Biogen-Idec Investigator, Principal Investigator — Biogen